CLINICAL TRIAL: NCT07033819
Title: A Single-arm, Prospective Clinical Study of Fluzoparib in Combination With Apatinib for Neoadjuvant Treatment of Homologous Recombination Deficiency Homologous Recombination Deficiency(HRD)-Positive Advanced Ovarian Cancer
Brief Title: Neoadjuvant Treatment of Ovarian Cancer With Fluazoparib in Combination With Apatinib
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/463-4743
Record Dates: First submitted 2025-04-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; neoadjuvant therapy; targeted therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Neoadjuvant Therapy; apatinib; Preoperative Period; Drug Therapy; Opiate Substitution Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant therapy (Experimental): Participants will receive neoadjuvant therapy with fluzoparib and apatinib for a total of three cycles (21 days per cycle).
  Interventions: Drug: Neoadjuvant therapy with fluazoparib in combination with apatinib; Procedure: Preoperative Period; Drug: Chemotherapy; Drug: Maintenance treatment

INTERVENTIONS:
Drug: Neoadjuvant therapy with fluazoparib in combination with apatinib — Neoadjuvant Treatment Period Furazopanib: 150 mg, twice daily, orally, either before or after meals. It is recommended to take it within 0.5 hours after breakfast and dinner. Continuous administration for 3 weeks constitutes one cycle, for a total of three cycles.
  Apatinib: 250 mg, once daily, orally, recommended to be taken within 0.5 hours after breakfast. Continuous administration for 3 weeks constitutes one cycle, for a total of three cycles.
  Other Names: Neoadjuvant therapy
Procedure: Preoperative Period — Discontinue Furazopanib 7 days before surgery. Discontinue Apatinib 14 days before surgery. The specific timing will be assessed by the investigator based on postoperative wound healing.
Drug: Chemotherapy — Postoperative Adjuvant Chemotherapy Period (≥4 cycles) Paclitaxel: 150-175 mg/m², intravenous infusion, every 3 weeks (Q3W). Carboplatin: AUC 4-5, intravenous infusion, every 3 weeks (Q3W).
Drug: Maintenance treatment — Maintenance Treatment Period Furazopanib: 150 mg, twice daily, orally. Continuous administration for 3 weeks constitutes one cycle.
  Apatinib: 250 mg, once daily, orally. Continuous administration for 3 weeks constitutes one cycle.
  Treatment will continue until disease progression, intolerable toxicity, or other reasons as specified in the protocol.

SUMMARY:
In this study, investigators propose to use fluzoparib and apatinib as neoadjuvant therapy for Homologous recombination deficiency （HRD）positive advanced ovarian cancer patients, aiming to explore the efficacy and safety of this 'de-chemotherapy' regimen as neoadjuvant therapy for advanced ovarian cancer, and to conduct genetically related subgroup analyses, to guide the precision therapy and provide a new therapeutic option for HRD-positive patients with advanced ovarian cancer. To provide a new treatment option In order to increase the R0 resection rate of surgery and reduce chemotherapy resistance, thus improving the prognosis and prolonging the survival of patients.

DETAILED DESCRIPTION:
This study is a single-arm, interventional, open-label, prospective clinical trial. Patients with advanced epithelial ovarian cancer (Federation of International of Gynecologists and Obstetricians，FIGO stage III-IV), who are not eligible for R0 resection or unable to tolerate surgery based on radiological assessment (Suidan score) or laparoscopic assessment (Fagotti score), and who are Homologous recombination deficiency （HRD）positive, will receive neoadjuvant therapy with fluzoparib and apatinib for three cycles (21 days per cycle). After neoadjuvant treatment, patients who achieve complete or partial response according to radiological assessment will proceed to the surgical treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer, with FIGO stage III-IV.
* Age between 18 and 70 years.
* Histopathological confirmation via laparoscopic biopsy or core needle biopsy indicating high-grade (or moderately/lowly differentiated) serous carcinoma, endometrioid carcinoma, fallopian tube cancer, or primary peritoneal cancer.
* Eastern Cooperative o ncology Group (ECOG) performance status of 0-1.
* Positive for homologous recombination deficiency (HRD) based on tissue or blood sample testing.
* Presence of at least one measurable lesion assessable by CT or MRI (RECIST v1.1).
* Ineligibility for primary debulking surgery due to inability to achieve R0 resection or intolerance to surgery, based on: Fagotti laparoscopic score ≥8. Upper abdominal CT score ≥3 when laparoscopic assessment is not feasible. Judgment criteria for surgery intolerance: BMI ≥40.0. Multiple chronic diseases. Malnutrition or hypoalbuminemia. Moderate to large volume ascites. Newly diagnosed venous thromboembolism.

ECOG performance status >2.

* Expected survival of >3 months.
* Adequate organ function, with laboratory results meeting the following criteria within 7 days prior to treatment initiation:

Hematological tests (no transfusions or hematopoietic growth factor use within 7 days prior to screening): Hemoglobin (Hb) ≥90 g/L. Absolute neutrophil count (ANC) ≥1.5×10⁹/L. Absolute lymphocyte count (LC) ≥0.5×10⁹/L. Platelet count (PLT) ≥100×10⁹/L. White blood cell count (WBC) ≥3.0×10⁹/L and ≤15×10⁹/L. Biochemical tests (no transfusions or albumin use within 7 days prior to screening): Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. Alkaline phosphatase (ALP) ≤2.5×ULN. Total bilirubin (TBIL) ≤1.5×ULN.

Serum creatinine (Cr) ≤1.5×ULN, with creatinine clearance (CrCL) ≥60 mL/min (Cockcroft-Gault formula). Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN, with international normalized ratio (INR) ≤1.5×ULN (not receiving anticoagulant therapy).

Urinalysis: Urine protein <2+; if urine protein ≥2+, then 24-hour urine protein quantification must show protein ≤1 g. 12-lead electrocardiogram (ECG): Fridericia-corrected QT interval (QTcF) <470 ms for females.

* Women of childbearing potential must have a negative serum or urine pregnancy test within one week prior to enrollment and must agree to use effective contraception during the study.
* Any prior chemotherapy-related toxicities must have resolved to ≤CTCAE Grade 1 or baseline, except for stable sensory neuropathy or alopecia of ≤CTCAE Grade 2.
* Voluntary participation in the study, with signed informed consent, good compliance, and willingness to participate in follow-up visits.

Exclusion Criteria:

* Hypersensitivity to the investigational drug or its excipients.
* Concurrent use of other neoadjuvant therapies for tumors during the study, including but not limited to chemotherapy, radiotherapy, immunotherapy, microbiological therapy, traditional Chinese medicine, or other experimental therapies.
* Inability to swallow oral medications, or presence of gastrointestinal diseases that may interfere with the absorption or metabolism of the study drug, such as uncontrollable nausea and vomiting, gastrointestinal obstruction, or malabsorption.
* Prior anti-cancer treatment for ovarian cancer.
* Previous treatment with known or potential PARP inhibitors or anti-angiogenic agents.
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids, or clinical manifestations of spinal cord compression.
* History of severe venous thromboembolism or pulmonary embolism.
* Receipt of other molecularly targeted therapies within 4 weeks prior to enrollment.
* Major surgery within one month prior to the start of the study, or not yet recovered from surgery.
* History of other malignancies within the past 3 years, except for adequately treated squamous cell carcinoma of the skin, basal cell carcinoma, ductal carcinoma in situ of the breast, or cervical carcinoma in situ.
* Prior or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Severe, uncontrolled medical conditions or investigator judgment that the participant is not suitable for the study, including but not limited to: active viral infections such as human immunodeficiency virus (HIV), hepatitis B, hepatitis C; severe cardiovascular disease, uncontrolled ventricular arrhythmias, myocardial infarction within the past 3 months; uncontrolled grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, or other psychiatric disorders affecting the ability to provide informed consent; uncontrolled hypertension; immunodeficiency (except splenectomy) or other diseases that the investigator deems may expose the patient to high-risk toxicity.
* Infection with human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis B, hepatitis C (positive for HCV antibody and HCV-RNA above the lower limit of detection of the assay), or co-infection with hepatitis B and C.
* Receipt of solid organ or hematopoietic stem cell transplantation during the study period (except for corneal transplantation).
* Current participation in another interventional clinical study, or receipt of other investigational drugs or devices within 4 weeks prior to the first dose; not fully recovered from toxicities and/or complications of any prior interventions (i.e., ≤Grade 1 or returned to baseline, excluding fatigue or alopecia).
* Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg despite optimal medical therapy).
* Abnormal coagulation function (INR >1.5 or prothrombin time (PT) >ULN + 4 seconds or APTT >1.5×ULN), history of bleeding tendency, or receiving thrombolytic or anticoagulant therapy.
* Urinalysis showing proteinuria ≥++, or confirmed 24-hour urine protein ≥1.0 g.
* History of substance abuse involving psychoactive drugs that cannot be discontinued, or participants with psychiatric disorders.
* History of hereditary or acquired bleeding disorders or coagulopathies (specific inclusion to be determined by the investigator).
* Concurrent use of strong CYP3A4 inhibitors (e.g., itraconazole, telithromycin, clarithromycin), moderate CYP3A4 inhibitors (e.g., ciprofloxacin, erythromycin, fluconazole), strong CYP3A4 inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampin), or moderate CYP3A4 inducers (e.g., bosentan, modafinil). A washout period of 5 weeks is required before study treatment for enzalutamide or phenobarbital, and 3 weeks for other drugs.
* History of stroke or transient ischemic attack within the past 6 months.
* Pregnant, breastfeeding, or planning to become pregnant during the study period (female participants).
* Other severe medical or psychiatric conditions or laboratory abnormalities that may increase the risk of participation, interfere with study treatment or outcomes, or any other situation deemed by the investigator as unsuitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | 4 months
  Proportion of patients with advanced epithelial ovarian cancer who are not R0 resectable at first diagnosis or who cannot tolerate surgery who undergo tumour cytoreduction to achieve R0 resection.

SECONDARY OUTCOMES:
Objective Remission Rate (ORR) | 24 months
  The proportion of patients whose tumor volume decreases by a predetermined amount and maintains this reduction for the minimum required duration. It is the sum of the complete response (CR) and partial response (PR) rates. In other words, ORR = CR + PR.
Progression-Free Survival (PFS) | 24 months
  The time from randomization until tumor progression (as defined by RECIST 1.1 criteria) or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | 24 months
  The percentage of evaluable patients who achieve a response (PR + CR) or stable disease (SD) after treatment. Simply put, DCR = CR + PR + SD, according to the RECIST criteria for at least 4 weeks.
Overall Survival (OS) | 36 months
  The time from randomization until death from any cause. For subjects who are lost to follow-up before death, the last follow-up time is usually counted as the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No